CLINICAL TRIAL: NCT00423631
Title: Internet-Enhanced Management of Fibromyalgia
Brief Title: Web-based Education to Enhance Fibromyalgia Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, David A. Williams, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAMD 17-002-0018, A-9356.1
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Fibromyalgia; Fibrositis
Keywords: Pain; Fibromyalgia; Internet
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care and Web (Experimental): Standard care plus a web site based on cognitive behavioral principals.
  Interventions: Behavioral: Standard care and web
- Standard Care (Active Comparator): Subject recieve standard care from their primary care provider.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Standard care and web — A static web site containing cognitive and behavioral self management instructions.
  Arms: Standard Care and Web
Behavioral: Standard Care — Standard care delivered by the primary care provider.
  Arms: Standard Care

SUMMARY:
Fibromyalgia (FMS) a condition marked by pain, fatigue, and memory complaints, is considered a chronic condition and is most commonly treated or managed using medications. Previous studies have found benefit in adding cognitive-behavioral therapy (CBT), a non-medication intervention, to standard care in order to obtain better outcomes in terms of improved functional status and symptom reduction. While the addition of CBT to standard care has been shown to be beneficial, it is not a form of therapy that is widely available to patients with FMS. CBT includes a variety of skills that can be taught to patients to help in the management of chronic illnesses. This protocol will examine the relative merits of providing these CBT skills to patients via an informational website. The website will contain the content of CBT, a social support capability, and data transfer capabilities. The addition of this website to standard care will be compared to standard care alone. This study is interested in assessing improvements in physical functional status, the symptoms of FMS, and the relative costs of the interventions as compared to the savings in health care utilization over a 6-month period.

Primary Hypothesis The primary hypothesis of this study is that the number of patients with fibromyalgia who are able to achieve clinically meaningful improvements in physical function will be greater when standard symptom-based pharmacological care is augmented by CBT skills delivered through an educational website.

Secondary Hypotheses

1. The proportion of patients with fibromyalgia who are able to achieve clinically meaningful improvements in symptoms of FMS such as pain, fatigue, and perceived cognitive difficulties will be greater when standard symptom-based pharmacological care is augmented by CBT skills delivered through an educational website
2. The proportion of patients with fibromyalgia who are able to achieve clinically meaningful improvements in mood and beliefs about pain will be greater when standard symptom-based pharmacological care is augmented by CBT skills delivered through an educational website

DETAILED DESCRIPTION:
Cognitive-Behavioral Therapy is a therapeutic approach that uses specific techniques to produce behavioral and cognitive change. CBT is not a singular approach to all problems; rather it is a set of techniques that can be tailored for specific problems. The techniques falling under the rubric of CBT have in common a scientific foundation based in learning and cognitive principles. The techniques used to change behavior are based on principles of classical and operant conditioning (e.g. extinction, positive and negative reinforcement, shaping, prompts), and observational learning. The techniques used to produce cognitive change are based largely on the development of problem solving skills and principles of attributional change (Craighead, Craighead, Kazdin, & Mahoney, 1994).

Cognitive behavioral therapy has been shown to be effective in the management of symptoms for a wide range of chronic medical illnesses (Compas, Haaga, Keefe, Leitenberg, & Williams, 1998; Emmelkamp & van Oppen, 1993; Gil et al., 1996)(1994; Emmelkamp et al., 1993; Turner & Romano, 1990; Gil et al., 1996; Keefe, 1996) including Fibromyalgia (Bradley, 1989; Nielson, Walker, & McCain, 1992; White & Nielson, 1995; Goldenberg, Kaplan, & Nadeau, 1994; Nielson et al., 1992; White et al., 1995; Goldenberg et al., 1994) and related conditions such as chronic fatigue syndrome (Sharpe et al., 1996; Deale, Chalder, Marks, & Wessely, 1997; Deale, Chalder, Marks, & Wessely, 1997). The rationale for using CBT with FMS stems from the assumption that pain and suffering is the result of a complex integration of pathophysiology, cognition, affect, and behavior (Keefe, 1996). Modification of any one of these four factors can positively or negatively impact the course of the persistent medical condition.

When applied to patients having fibromyalgia, CBT has been shown to be associated with both short-term (3 weeks) and long-term (30 months) improvements in pain, distress, and perceived control over pain (Nielson et al., 1992; White et al., 1995; White et al., 1995). Several other investigations of CBT have demonstrated improvements in depression, pain behaviors, and tenderness (Nicassio et al., 1997), as well as knowledge of fibromyalgia and coping with pain (Vlaeyen et al., 1996). While the latter two studies did not demonstrate a superiority of CBT over educational approaches, a meta-analytic review concluded that psychological interventions for fibromyalgia in general produced effect sizes that exceeded those of physical therapy or pharmacological interventions for outcomes such as symptoms, mental health, and physical functioning (Rossy et al., 1999). The latter outcome, a sustained improvement in physical functioning, was the most difficult outcome to achieve for patients with fibromyalgia using any form of intervention. One recent study however demonstrated that 1-year sustained improvements in physical functional status were three times more likely in patients that attended a brief course of CBT than if they received only symptom-based pharmacological care (Williams, 2002).

New Advances in CBT Delivery Despite the demonstrated effectiveness of combining pharmacological interventions with CBT, integration of CBT into mainstream clinical practice for FMS has been slow. Barriers have not been due to lack of demonstrated efficacy, but rather to economic and administrative issues such as the lack of CPT codes for applying a psychological intervention for a physical illness, difficulties administering a time-intensive psychological intervention to populations that must travel long distances each week to obtain the intervention, and the lack of sufficient numbers of trained professionals to deliver the intervention on a large scale (Muehrer, 2000).

A current technology, Internet websites, has been implemented in an effort to overcome some of the barriers that have prevented the delivery of clinical services to FMS populations.

Healthcare Websites E-learning, the use of a website for education without the use of a live instructor, has become a popular method for educating the lay-public, for offering classes for credit and for continuing education online, and for training employees new job skills. Numerous websites exist that purport to improve health. Some of these sites simply provide information about illness, others provide interactive preprogrammed advice, and some send tailored health messages to patients.

The current study will seek to evaluate the effectiveness of using traditional standard care with standard care plus Internet web-based educational programming. This will be one of the largest randomized controlled trials to use web-based learning and should help to identify the feasibility of using this modality to augment standard care for the FMS community.

ELIGIBILITY:
SUBJECTS WILL NEED TO COME TO SIOUX FALLS FOR THE STUDY VISITS.

The study sample will be drawn from a population of individuals diagnosed with fibromyalgia in a five state region consisting of North and South Dakota, Iowa, Minnesota, and Nebraska.

Subjects will be recruited into the study by practicing physicians either at the main hospital in Sioux Falls or in any of 15 affiliated rural clinic study sites. In order to be included in the study, potential subjects must meet the study inclusion and exclusion criteria.

Inclusion Criteria:

1. Ability to travel to Sioux Falls, SD for study visits.
2. All subjects must fulfill the diagnostic criteria for fibromyalgia as established by the American College of Rheumatology (ACR) in 1990 (Wolfe et al., 1990)
3. Be 18 years of age
4. All subjects must have been in standard medical care with a physician for at least 3 months.
5. Subjects must have a home computer or access to a computer with the following features:

   * An Internet browser that is Internet Explorer version 5.0 or higher.
   * Printer
   * Speakers or headphones
   * Ability to use e-mail and access to the Internet
6. Subjects must be able to perform the following screening test designed to assess computer ability:

   * Go to a webpage Log in to a website
   * Click on an icon
   * Click on a radio button to answer a multiple choice question
   * Fill a name into a text box
   * Click on a submit button
   * Print a document

Exclusion Criteria:

Subjects will be excluded from participation if they have any of the following:

1. A severe physical impairment that precludes receiving/using the website or using the CBT skills contained on the website (e.g. complete blindness)
2. Co-morbid medical illnesses capable of causing a worsening of physical functional status independent of fibromyalgia (e.g. morbid obesity, autoimmune diseases,) cardiopulmonary disorders (e.g. angina, congestive heart failure, COPD, chronic asthma), uncontrolled endocrine or allergic disorders (e.g. thyroid dysfunction, Type I diabetes), and malignancy within 2 years.
3. Any present psychiatric disorder involving a history of psychosis (e.g. schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder etc.), current suicide risk or attempt within 2 years of the study, or substance abuse within 2 years. Note: Subjects with mood disorders will not be excluded.
4. Prior face to face CBT for pain management.
5. Receiving or applying for or considering seeking disability payments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Clinically meaningful improvements in physical function (as measured by the SF-36). | baseline to 6 months
Clinically meaningful improvements in symptoms of FMS such as pain, fatigue, and perceived cognitive difficulties (as measured by the McGill, MFI and MASQ). | baseline to 6 months
Clinically meaningful improvements in mood and beliefs about pain (as measured by the CES-D, STPI, CSQ and BPCQ) | baseline to 6 months

SECONDARY OUTCOMES:
To determine whether treatment adherence is superior in one of the treatment arms of the study, and whether adherence is related to improved outcomes. | baseline to 6 months
To determine whether treatment satisfaction is superior in one of the treatment arms of the study, and whether that satisfaction is related to improved outcomes | Baseline to 6 months
To determine post hoc, the characteristics of the individuals that achieved treatment success versus those that did not, to better identify the factors that contribute to positive outcomes in this spectrum of illness. | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David A Williams, PhD, Principal Investigator — University of Michigan
Locations (1):
- Avera Research Institute, Sioux Falls, South Dakota, United States

REFERENCES:
- [Background] Fukuda K, Nisenbaum R, Stewart G, Thompson WW, Robin L, Washko RM, Noah DL, Barrett DH, Randall B, Herwaldt BL, Mawle AC, Reeves WC. Chronic multisymptom illness affecting Air Force veterans of the Gulf War. JAMA. 1998 Sep 16;280(11):981-8. doi: 10.1001/jama.280.11.981. PMID 9749480
- [Background] Clauw DJ, Chrousos GP. Chronic pain and fatigue syndromes: overlapping clinical and neuroendocrine features and potential pathogenic mechanisms. Neuroimmunomodulation. 1997 May-Jun;4(3):134-53. doi: 10.1159/000097332. PMID 9500148
- [Background] Clauw DJ. Fibromyalgia: more than just a musculoskeletal disease. Am Fam Physician. 1995 Sep 1;52(3):843-51, 853-4. PMID 7653424
- [Background] Crofford LJ, Engleberg NC, Demitrack MA. Neurohormonal perturbations in fibromyalgia. Baillieres Clin Rheumatol. 1996 May;10(2):365-78. doi: 10.1016/s0950-3579(96)80022-7. PMID 8911654
- [Background] Wolfe F, Ross K, Anderson J, Russell IJ, Hebert L. The prevalence and characteristics of fibromyalgia in the general population. Arthritis Rheum. 1995 Jan;38(1):19-28. doi: 10.1002/art.1780380104. PMID 7818567
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Yunus MB. Towards a model of pathophysiology of fibromyalgia: aberrant central pain mechanisms with peripheral modulation. J Rheumatol. 1992 Jun;19(6):846-50. No abstract available. PMID 1404119
- [Background] Carette S, Bell MJ, Reynolds WJ, Haraoui B, McCain GA, Bykerk VP, Edworthy SM, Baron M, Koehler BE, Fam AG, et al. Comparison of amitriptyline, cyclobenzaprine, and placebo in the treatment of fibromyalgia. A randomized, double-blind clinical trial. Arthritis Rheum. 1994 Jan;37(1):32-40. doi: 10.1002/art.1780370106. PMID 8129762
- [Background] Godfrey RG. A guide to the understanding and use of tricyclic antidepressants in the overall management of fibromyalgia and other chronic pain syndromes. Arch Intern Med. 1996 May 27;156(10):1047-52. PMID 8638990
- [Background] Compas BE, Haaga DA, Keefe FJ, Leitenberg H, Williams DA. Sampling of empirically supported psychological treatments from health psychology: smoking, chronic pain, cancer, and bulimia nervosa. J Consult Clin Psychol. 1998 Feb;66(1):89-112. doi: 10.1037//0022-006x.66.1.89. PMID 9489263
- [Background] Emmelkamp PM, van Oppen P. Cognitive interventions in behavioral medicine. Psychother Psychosom. 1993;59(3-4):116-30. doi: 10.1159/000288656. PMID 8416088
- [Background] Gil KM, Wilson JJ, Edens JL, Webster DA, Abrams MA, Orringer E, Grant M, Clark WC, Janal MN. Effects of cognitive coping skills training on coping strategies and experimental pain sensitivity in African American adults with sickle cell disease. Health Psychol. 1996 Jan;15(1):3-10. doi: 10.1037//0278-6133.15.1.3. PMID 8788535
- [Background] The Persian Gulf experience and health. NIH Technology Assessment Workshop Panel. JAMA. 1994 Aug 3;272(5):391-6. No abstract available. PMID 8028172
- [Background] Bradley LA. Cognitive-behavioral therapy for primary fibromyalgia. J Rheumatol Suppl. 1989 Nov;19:131-6. PMID 2691672
- [Background] White KP, Nielson WR. Cognitive behavioral treatment of fibromyalgia syndrome: a followup assessment. J Rheumatol. 1995 Apr;22(4):717-21. PMID 7791170
- [Background] Sharpe M, Hawton K, Simkin S, Surawy C, Hackmann A, Klimes I, Peto T, Warrell D, Seagroatt V. Cognitive behaviour therapy for the chronic fatigue syndrome: a randomized controlled trial. BMJ. 1996 Jan 6;312(7022):22-6. doi: 10.1136/bmj.312.7022.22. PMID 8555852
- [Background] Deale A, Chalder T, Marks I, Wessely S. Cognitive behavior therapy for chronic fatigue syndrome: a randomized controlled trial. Am J Psychiatry. 1997 Mar;154(3):408-14. doi: 10.1176/ajp.154.3.408. PMID 9054791
- [Background] Nicassio PM, Radojevic V, Weisman MH, Schuman C, Kim J, Schoenfeld-Smith K, Krall T. A comparison of behavioral and educational interventions for fibromyalgia. J Rheumatol. 1997 Oct;24(10):2000-7. PMID 9330945
- [Background] Vlaeyen JW, Teeken-Gruben NJ, Goossens ME, Rutten-van Molken MP, Pelt RA, van Eek H, Heuts PH. Cognitive-educational treatment of fibromyalgia: a randomized clinical trial. I. Clinical effects. J Rheumatol. 1996 Jul;23(7):1237-45. PMID 8823699
- [Background] Rossy LA, Buckelew SP, Dorr N, Hagglund KJ, Thayer JF, McIntosh MJ, Hewett JE, Johnson JC. A meta-analysis of fibromyalgia treatment interventions. Ann Behav Med. 1999 Spring;21(2):180-91. doi: 10.1007/BF02908299. PMID 10499139
- [Background] Williams DA, Cary MA, Groner KH, Chaplin W, Glazer LJ, Rodriguez AM, Clauw DJ. Improving physical functional status in patients with fibromyalgia: a brief cognitive behavioral intervention. J Rheumatol. 2002 Jun;29(6):1280-6. PMID 12064847
- [Background] Muehrer P. Research on adherence, behavior change, and mental health: a workshop overview. Health Psychol. 2000 May;19(3):304-7. doi: 10.1037//0278-6133.19.3.304. PMID 10868776
- [Background] Horowitz LM, Rosenberg SE, Baer BA, Ureno G, Villasenor VS. Inventory of interpersonal problems: psychometric properties and clinical applications. J Consult Clin Psychol. 1988 Dec;56(6):885-92. doi: 10.1037//0022-006x.56.6.885. No abstract available. PMID 3204198
- [Background] Ware JE Jr, Bayliss MS, Rogers WH, Kosinski M, Tarlov AR. Differences in 4-year health outcomes for elderly and poor, chronically ill patients treated in HMO and fee-for-service systems. Results from the Medical Outcomes Study. JAMA. 1996 Oct 2;276(13):1039-47. PMID 8847764
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Schluederberg A, Straus SE, Peterson P, Blumenthal S, Komaroff AL, Spring SB, Landay A, Buchwald D. NIH conference. Chronic fatigue syndrome research. Definition and medical outcome assessment. Ann Intern Med. 1992 Aug 15;117(4):325-31. doi: 10.7326/0003-4819-117-4-325. PMID 1322076
- [Background] Geisser ME, Robinson ME, Keefe FJ, Weiner ML. Catastrophizing, depression and the sensory, affective and evaluative aspects of chronic pain. Pain. 1994 Oct;59(1):79-83. doi: 10.1016/0304-3959(94)90050-7. PMID 7854806
- [Background] Sullivan MJ, D'Eon JL. Relation between catastrophizing and depression in chronic pain patients. J Abnorm Psychol. 1990 Aug;99(3):260-3. doi: 10.1037//0021-843x.99.3.260. PMID 2145334
- [Background] Keefe FJ, Brown GK, Wallston KA, Caldwell DS. Coping with rheumatoid arthritis pain: catastrophizing as a maladaptive strategy. Pain. 1989 Apr;37(1):51-56. doi: 10.1016/0304-3959(89)90152-8. PMID 2726278
- [Background] Jensen MP, Turner JA, Romano JM, Karoly P. Coping with chronic pain: a critical review of the literature. Pain. 1991 Dec;47(3):249-283. doi: 10.1016/0304-3959(91)90216-K. PMID 1784498
- [Background] Lacker JM, Carosella AM, Feuerstein M. Pain expectancies, pain, and functional self-efficacy expectancies as determinants of disability in patients with chronic low back disorders. J Consult Clin Psychol. 1996 Feb;64(1):212-20. doi: 10.1037//0022-006x.64.1.212. PMID 8907101
- [Background] Williams DA, Thorn BE. An empirical assessment of pain beliefs. Pain. 1989 Mar;36(3):351-358. doi: 10.1016/0304-3959(89)90095-X. PMID 2710564
- [Background] Jensen MP, Turner JA, Romano JM, Lawler BK. Relationship of pain-specific beliefs to chronic pain adjustment. Pain. 1994 Jun;57(3):301-309. doi: 10.1016/0304-3959(94)90005-1. PMID 7936708
- [Background] Rosenstiel AK, Keefe FJ. The use of coping strategies in chronic low back pain patients: relationship to patient characteristics and current adjustment. Pain. 1983 Sep;17(1):33-44. doi: 10.1016/0304-3959(83)90125-2. PMID 6226916
- [Background] Keefe FJ, Crisson J, Urban BJ, Williams DA. Analyzing chronic low back pain: the relative contribution of pain coping strategies. Pain. 1990 Mar;40(3):293-301. doi: 10.1016/0304-3959(90)91126-4. PMID 2139204
- [Background] Keefe FJ, Caldwell DS, Martinez S, Nunley J, Beckham J, Williams DA. Analyzing pain in rheumatoid arthritis patients. Pain coping strategies in patients who have had knee replacement surgery. Pain. 1991 Aug;46(2):153-160. doi: 10.1016/0304-3959(91)90070-E. PMID 1749638
- [Background] Nielson WR, Walker C, McCain GA. Cognitive behavioral treatment of fibromyalgia syndrome: preliminary findings. J Rheumatol. 1992 Jan;19(1):98-103. PMID 1556709
- [Background] Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID 2912463
- [Background] Williams DA, Robinson ME, Geisser ME. Pain beliefs: assessment and utility. Pain. 1994 Oct;59(1):71-78. doi: 10.1016/0304-3959(94)90049-3. PMID 7854805
- [Background] Lipchik GL, Milles K, Covington EC. The effects of multidisciplinary pain management treatment on locus of control and pain beliefs in chronic non-terminal pain. Clin J Pain. 1993 Mar;9(1):49-57. doi: 10.1097/00002508-199303000-00007. PMID 8477140
- [Background] Jensen MP, Keefe FJ, Lefebvre JC, Romano JM, Turner JA. One- and two-item measures of pain beliefs and coping strategies. Pain. 2003 Aug;104(3):453-469. doi: 10.1016/S0304-3959(03)00076-9. PMID 12927618
- [Background] Jensen MP, Turner JA, Romano JM, Strom SE. The Chronic Pain Coping Inventory: development and preliminary validation. Pain. 1995 Feb;60(2):203-216. doi: 10.1016/0304-3959(94)00118-X. PMID 7784106
- [Background] Nguyen TD, Attkisson CC, Stegner BL. Assessment of patient satisfaction: development and refinement of a service evaluation questionnaire. Eval Program Plann. 1983;6(3-4):299-313. doi: 10.1016/0149-7189(83)90010-1. PMID 10267258
- [Background] Walters SJ, Brazier JE. What is the relationship between the minimally important difference and health state utility values? The case of the SF-6D. Health Qual Life Outcomes. 2003 Apr 11;1:4. doi: 10.1186/1477-7525-1-4. PMID 12737635
- [Background] Lachin JM. Introduction to sample size determination and power analysis for clinical trials. Control Clin Trials. 1981 Jun;2(2):93-113. doi: 10.1016/0197-2456(81)90001-5. PMID 7273794